CLINICAL TRIAL: NCT05467696
Title: A Phase 1 Open-Label, Two-Period, Two-Treatment, Crossover Study of the Effect of Food on the Bioavailability of the To-Be-Marketed Formulation of CTP-543 in Healthy Volunteers
Brief Title: Study of the Effect of Food on the Bioavailability of the To-Be-Marketed Formulation of CTP-543 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CP543.1011
Record Dates: First submitted 2022-06-30; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Health Volunteers
Keywords: CTP-543

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 Fed:Fasted (Experimental): Period 1: CTP-543 12 mg fed Period 2: CTP-543 12 mg fasted
  Interventions: Drug: CTP-543
- Sequence 2 Fasted:Fed (Experimental): Period 1: CTP-543 12 mg fasted Period 2: CTP-543 12 mg fed
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — For each period, subjects will be dosed with CTP-543 12 mg (1 x 12 mg tablet)

SUMMARY:
This is an open-label, single-dose, two period crossover study to evaluate the effect of food on the bioavailability of the To-Be-Marketed Formulation of CTP-543 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18-60 years of age, inclusive
* Nonsmoker who has not used nicotine containing products for at least 3 months
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs
* If of reproductive age, willing and able to use a medically highly effective form of birth control 4 weeks prior to first dose, during the study and for 30 days following last dose of study medication
* Capable of giving informed consent and complying with study procedures.

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History of any illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study
* History or presence of alcohol or drug abuse within the past 2 years
* Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
* History of prolonged QT syndrome or a QTc interval with Fridericia's correction (QTcF) > 450 msec for males or QTcF > 470 msec for females
* Abnormal liver function at screening
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug
* Positive results for coronavirus infection (COVID-19) at screening or check-in (Day -1)
* Positive drug or alcohol results at screening
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Participation in another clinical study within 30 days prior to, and 30 days after the first dosing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-06-26 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Bioavailability and Pharmacokinetic Profile of CTP-543: Cmax | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Maximum observed concentration
Bioavailability and Pharmacokinetic Profile of CTP-543: Tmax | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Time to reach maximum observed concentration
Bioavailability and Pharmacokinetic Profile of CTP-543: AUC(0-Tlast) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Area under the concentration-time curve from time 0 to the time of the last observed/measured non-zero concentration
Bioavailability and Pharmacokinetic Profile of CTP-543: AUC(0-inf) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Area under the concentration-time curve from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Pharmacokinetic Profile of major metabolites: Cmax | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Maximum observed concentration
Pharmacokinetic Profile of major metabolites: Tmax | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Time to reach maximum observed concentration
Pharmacokinetic Profile of major metabolites: AUC(0-Tlast) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Area under the concentration-time curve from time 0 to the time of the last observed/measured non-zero concentration
Pharmacokinetic Profile of major metabolites: AUC(0-inf) | 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose and Day 6/discharge
  Area under the concentration-time curve from time 0 extrapolated to infinity
Assessment of Safety and Tolerability following administration of CTP-543 | Screening through 7 to 10 days after final dose administration
  Number of adverse events including abnormal clinical laboratory findings, abnormal physical examinations, abnormal ECGs and abnormal vital signs tabulated for each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States